CLINICAL TRIAL: NCT04072913
Title: Involvement of Matrix Metalloproteinases and Association With the Expression of Human Papillomavirus in Dysplasias and Cancers of the Cervix
Brief Title: Matrix Metalloproteinases and Human Papillomavirus in Dysplasias and Cancers of the Cervix
Acronym: MMP-HPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2007/08
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Papillomavirus Infections; Dysplasia; Cervix Cancer
Keywords: Matrix metalloproteinases
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms | interventions — Biopsy; Vaginal Smears

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (Other): Study of the expression of matrix metalloproteinases and their tissue inhibitors
  Interventions: Other: Vaginal samples (biopsies + vaginal smear)
- Low grade lesion group (Other): Study of the expression of matrix metalloproteinases and their tissue inhibitors
  Interventions: Other: Vaginal samples (biopsies + vaginal smear)
- High grade lesions group (Other): Study of the expression of matrix metalloproteinases and their tissue inhibitors
  Interventions: Other: Vaginal samples (biopsies + vaginal smear)
- Cancer group (Other): Study of the expression of matrix metalloproteinases and their tissue inhibitors
  Interventions: Other: Vaginal samples (biopsies + vaginal smear)

INTERVENTIONS:
Other: Vaginal samples (biopsies + vaginal smear) — Two types of samples are envisaged: tissue (large biopsies, coin of conization or hysterectomy) to affirm the diagnosis and detect the matrix metalloproteinases and their tissue inhibitors by immunohistochemistry; cell sample (monolayer smear type) to evaluate the expression of oncogenic Human papillomavirus.

SUMMARY:
This study aims to compare the expression of matrix metalloproteinases and their tissue inhibitors between 4 groups of patients defined according to the severity of the cervical lesion.

DETAILED DESCRIPTION:
Cervical cancer is the second most common cancer among European women under 45 years old. It is secondary to cervical dysplasia induced by persistent human papillomavirus infection. The involvement of matrix metalloproteinases in carcinogenesis of the cervix is real, but their expressions vary according to the published series. An association between the expression of MMPs and that of the human papillomavirus deserves to be explored, as this can have a prognostic influence in the case of gradual expression demonstrated in the development of (pre) cancerous lesions of the cervix.

This study aims to compare the expression of matrix metalloproteinases and their tissue inhibitors between 4 groups of patients defined according to the severity of the cervical lesion.

ELIGIBILITY:
Inclusion Criteria:

For control group:

* Age between 20 and 65 years
* Patients hospitalized for partial or total removal of the cervix
* Absence of cervical lesion observed on biopsy or hysterectomy
* Free, informed and written consent, dated and signed by the patient and the investigator (at the latest before any examination required by the study)
* Affiliate or beneficiary of a social security scheme

For dysplasia and cancer group:

* Age between 20 and 65 years
* Cervical Intraepithelial Neoplasia or previously untreated cervical cancer
* Free, informed and written consent, dated and signed by the patient and the investigator (at the latest before any examination required by the study)
* Affiliate or beneficiary of a social security scheme

Exclusion Criteria:

For control group:

* History of laser or conisation
* Known antecedent of HIV infection
* Congenital or acquired immunodepression
* Long-term treatment with corticosteroids or immunosuppressants
* Persons placed under the protection of justice

For dysplasia and cancer group:

* History of laser or conisation
* Pre-treatment of invasive cancers by radiotherapy or chemotherapy
* Known antecedent of HIV infection
* Congenital or acquired immunodepression
* Long-term treatment with corticosteroids or immunosuppressants
* Persons placed under the protection of justice

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study on cervix
Enrollment: 216 (Actual)
Dates: Start 2007-10-10 (Actual); Primary Completion 2011-01-31 (Actual); Study Completion 2011-01-31 (Actual)

PRIMARY OUTCOMES:
Immunohistochemical score of expressions of matrix metalloproteinases | At the screening
  The immunohistochemical score is the modified HScore, also called Quickscore. It is calculated by multiplying the percentage of cells that are marked (from 0 to 100) by intensity (from 0 to 3). The total score is between 0 and 300. This score will be defined on normal, tumoral and stromal cells according to the analyzed tissue (normal, dysplasias or cancer)
Immunohistochemical score of expressions of matrix metalloproteinases inhibitors | At the screening
  The immunohistochemical score is the modified HScore, also called Quickscore. It is calculated by multiplying the percentage of cells that are marked (from 0 to 100) by intensity (from 0 to 3). The total score is between 0 and 300. This score will be defined on normal, tumoral and stromal cells according to the analyzed tissue (normal, dysplasias or cancer)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc BRUN, Dr, Principal Investigator — University Hospital, Bordeaux

IPD SHARING:
Plan to Share IPD: No